CLINICAL TRIAL: NCT02101593
Title: A Phase 1 Study of ADI PEG 20 Plus Sorafenib in Subjects With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Ph 1 Trial of ADI PEG 20 Plus Sorafenib to Treat Patients With Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-005
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental)
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20
  Other Names: arginine deiminase formulated with polyethylene glycol

SUMMARY:
Assessment of safety and tolerability of ADI-PEG 20 in combination with sorafenib in advanced Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of HCC confirmed histologically.
2. HCC tissue either from an archived specimen or from a new biopsy of sufficient amount and quality should be available for IHC determination of ASS status, and other biomarkers, to be performed retrospectively. Subjects with no tissue available would require a biopsy.
3. No prior treatment with systemic chemotherapy (except as noted in exclusion criteria # 10).
4. Measurable disease using RECIST 1.1 criteria (Appendix A). At least 1 measurable lesion must be present. Subjects who have received local-regional therapy such as (but not limited to) chemoembolization, embolization, cryoablation, hepatic artery therapy, percutaneous ethanol injection, radiation therapy, radiofrequency ablation or surgery are eligible, provided that they have either a target lesion which has not been treated with local therapy and/or the target lesion(s) within the field of the local regional therapy has shown an increase of ≥ 20% in size. Local-regional therapy must be completed at least 4 weeks prior to the baseline CT scan. Local therapies including chemoembolization do not count as prior systemic therapy.
5. Cirrhotic status of Child-Pugh grade A. Child-Pugh status should be determined based on clinical findings and laboratory data during the screening period (Appendix B). Subjects on anti-coagulants are to receive 1 point for their INR status, as they are presumed to have a <1.7 baseline PT/INR.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Appendix C).
7. Expected survival of at least 3 months.
8. Age ≥ 18 years.

Exclusion Criteria:

1. Candidate for potential curative therapies (i.e., resection or transplantation).
2. Prior allograft transplantation including liver transplantation.
3. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
4. Pregnancy or lactation.
5. Expected non-compliance.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV; Appendix D), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements.
7. Subjects who have not fully recovered from toxicities associated with previous HCC loco-regional therapies.
8. Subjects with history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current HCC diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of ADI-PEG 20 in combination with sorafenib in advanced HCC | course of study - 1 year expected

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center (MSKCC)
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington